CLINICAL TRIAL: NCT02376985
Title: Evaluation of Oral Care to Prevent Oral Mucositis in Estrogen Receptor Positive Metastatic Breast Cancer Patients Treated With Everolimus: Phase III Randomized Control Trial
Brief Title: Evaluation of Oral Care to Prevent Oral Mucositis in ER Positive MBC Patients Treated With Everolimus: Phase 3 RCT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Comprehensive Support Project for Oncology Research (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Oral Care-BC
Record Dates: First submitted 2015-02-26; First posted 2015-03-03 (Estimated); Last update posted 2019-10-21 (Actual); Status verified 2019-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Therapeutics; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Brushing instruction group (Placebo Comparator): Drug: Everolimus and Exemestane Everolimus, 10 mg/day Exemestane, 25 mg/day Administration on consecutive days once daily after breakfast until tumor progression or for a minimum 8 weeks.
  Oral treatment:
  Brushing and gargling with saline after every meal (initially instructed by a dental/oral surgeon).
  Interventions: Drug: Everolimus
- Dental oral management group (Experimental): Drug: Everolimus and Exemestane Everolimus, 10 mg/day Exemestane, 25 mg/day Administration on consecutive days once daily after breakfast until tumor progression or for a minimum 8 weeks.
  Oral treatment:
  Scaling and enamel polishing will be performed by a dental and oral surgeon or dental hygienist before everolimus treatment, and once weekly after everolimus treatment.
  Brushing and gargling with Neostelin Green 0.2% mouthwash solution after every meal (initially instructed by a dental/oral surgeon).
  Interventions: Procedure: Oral management; Drug: Everolimus

INTERVENTIONS:
Procedure: Oral management
  Arms: Dental oral management group
Drug: Everolimus

SUMMARY:
To examine whether the occurrence of oral mucositis can be reduced by dental oral management in patients by comparing the use of dental oral management through instruction by dental and oral surgeons (dental oral management group) and an observation group (brushing instruction only group) in a randomized, controlled study in females that are using everolimus for estrogen receptor-positive, hormone therapy-resistant refractory breast cancer.

DETAILED DESCRIPTION:
To examine whether the occurrence of oral mucositis can be reduced by dental oral management in patients by comparing the use of dental oral management through instruction by dental surgeons or oral surgeons (hereafter referred to as, "dental and oral surgeons") and an observation group in a randomized, controlled study in females that are using everolimus for estrogen receptor-positive, hormone therapy-resistant refractory breast cancer.

The objectives of this study are as described below.

1. To examine whether the occurrence of oral mucositis can be reduced by implementing dental oral management prior to everolimus treatment.
2. To examine whether the frequency and duration of oral mucositis can be reduced and reductions in the dose of everolimus can be reduced by implementing dental oral management prior to everolimus treatment.
3. To examine whether treatment of oral mucositis of over Grade 1 with dexaltin ointment as dental oral management can reduce the occurrence of Grade 2 oral mucositis.
4. To evaluate the health-related quality of life (HRQOL) in a group that implements dental oral management prior to everolimus treatment and a group that does not.
5. To establish and strengthen cooperation and organize and expand and information distribution network through the participation of oncologists and specialists in breast cancer treatment (hereafter referred to as, "oncologists") and dental and oral surgeons in clinical studies.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients with a histological diagnosis of breast cancer (regardless of histological subtype of breast cancer).
2. Diagnosis of metastatic or recurrent breast cancer satisfies either of the below.

   1. Distant metastasis present that is inoperable at time of first examination (Stage IV, 3.1 Clinical stage classification)
   2. Progression of distant metastasis or recurrence of breast cancer after treatment (after surgery and after treatments prior to and after surgery)
3. Histologically confirmed diagnosis of ER-positive breast cancer
4. Postmenopause
5. Any of the below conditions indicating resistance to aromatase inhibitor therapy. The aromatase inhibitor therapy need not be the most recent therapy.

   1. Recurrence during ongoing adjuvant therapy with an aromatase inhibitor, or recurrence within 12 months after adjuvant therapy with an aromatase inhibitor
   2. Progression during ongoing aromatase inhibitor therapy for advanced breast cancer, or progression within 1 month after ending aromatase inhibitor therapy
6. Any number of chemotherapy (anti-neoplastic drugs) are allowed since diagnosis of metastatic or recurrent breast cancer
7. Aged ≥20 years
8. PS of 0-1. (ECOG scale).
9. Previous treatment (including adjuvant therapy) satisfies all the conditions below.

   1. Hormone therapy: At least 7 days have elapsed from the last administration of hormonal therapy.
   2. Radiotherapy: At least 14 days have elapsed from the last irradiation.
10. Organ function (within 4 weeks before enrollment) satisfies all the conditions below.

    1. Neutrophil count (band cells + segmented cells) of ≥1,500/mm3, or white blood cell count of ≥3,000/mm3
    2. Platelet count of ≥100,000/mm3
    3. Total bilirubin of ≤2.5 × ULN
    4. AST (GOT) and ALT (GPT) of ≤2.5 × ULN
    5. Serum creatinine of ≤1.5 × ULN
11. Cardiac function satisfies either of the below.

    1. No cardiac disorder: No fatigue, palpitation, shortness of breath, or anginal pain during everyday activities as confirmed by interview.
    2. Has a cardiac disorder that does not limit movement, patient is confirmed to experience no fatigue, palpitation, shortness of breath, or anginal pain during everyday activities, and this health status is deemed to be maintained during treatment.
12. Informed consent is obtainable from the subject herself in documented form using the Consent Form.

Exclusion Criteria:

1. Edentulous jaw (in both upper and lower jaws)
2. Occurrence of oral mucositis within 1 month prior to randomization
3. Chemotherapy used within 1 month prior to randomization
4. Exemestane monotherapy (this exclusion criterion is not met if ≥3 months has elapsed since the last exemestane treatment) as most recent therapy
5. Previous mTOR inhibitor treatment (everolimus, etc.)
6. Interstitial pneumonia or pulmonary fibrosis.
7. Received drug treatment known to have a strong inhibitory or inductive effect on the cytochrome P450 (CYP) 3A isozymes (rifabutin, rifampicin, clarithromycin, ketoconazole, itraconazole, voriconazole, ritonavir, telithromycin) (See Table 4.1.2.1 and 4.1.2.2 for lists of prohibited concomitant drugs).
8. Positive result of HBs antigen, HBc antibody and/or HBs antibody.
9. HCV infection or a history of HCV infection.
10. History of hypersensitivity to a protocol treatment drug or a vehicle in the drug preparation.
11. Multiple active cancers (homochronous multiple cancers, or heterochronous multiple cancers with a cancer-free period of less than 5 years prior to randomization).

    Carcinoma in situ deemed to be cured by local treatment (lesions that are intraepithelial carcinoma or mucosal cancer) is not included as an active multiple cancer.
12. Overexpression of HER2 (Her2/neu, Erb B2), and the condition is considered to be indicated for trastuzumab (herceptin®) treatment (when the state of HER2 expression is unknown, the patient is not excluded, but is treated as eligible).

    In other words, patients that satisfy any of the below conditions will be excluded.

    At either the primary or the metastatic lesion:
    1. Strongly positive, "3+" by HER2 IHC.
    2. Positive "+" by FISH
13. Brain metastasis that requires treatment for intracranial hypertension or emergency irradiation of the brain.
14. Extensive liver metastasis, or lymphangitic lung metastasis with accompanying dyspnea.
15. Pleural effusion, ascites, or pericardial effusion that requires emergency treatment.
16. Concurrent and active infectious disease.
17. With uncontrolled diabetes mellitus or currently receiving insulin therapy.
18. Difficulty to participate in this study due to mental illness or psychiatric symptoms.
19. With another reasons recognized as inadequate to participate in this study by doctors.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2015-03-26 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-10-16 (Actual)

PRIMARY OUTCOMES:
Incidence of oral mucositis (Over Grade 1) after everolimus treatment | Patients are followed up for 8 weeks after initial enrollment
  Incidence of oral mucositis in Grade 1 or more, is evaluated by an oncologist.

SECONDARY OUTCOMES:
Incidence of oral mucositis (Over Grade 2) | Patients are followed up for 8 weeks after initial enrollment
  Incidence of oral mucositis in Grade 2 or more, is evaluated by an oncologist.
Incidence of oral mucositis (Over Grade 3) | Patients are followed up for 8 weeks after initial enrollment
  Incidence of oral mucositis in Grade 3 or more, is evaluated by an oncologist.
Incidence of oral mucositis (Over Grade 1) | Patients are followed up for 8 weeks after initial enrollment
  Incidence of oral mucositis in Grade 1 or more, is evaluated by a dental and oral surgeon
Incidence of oral mucositis (Over Grade 2) | Patients are followed up for 8 weeks after initial enrollment
  Incidence of oral mucositis in Grade 2 or more, is evaluated by a dental and oral surgeon
Incidence of oral mucositis (Over Grade 3) | Patients are followed up for 8 weeks after initial enrollment
  Incidence of oral mucositis in Grade 3 or more, is evaluated by a dental and oral surgeon
Time to the onset of oral mucositis | Patients are followed up for 8 weeks after initial enrollment
  Time to the onset of mucositis is evaluated by an oncologist or a dental/oral surgeon
Duration of each Grade of oral mucositis | Patients are followed up for 8 weeks after initial enrollment
  Duration of each Grade of mucositis is evaluated by an oncologist or a dental/oral surgeon, respectively
Each ratio of patients in suspension, or dose-reduction of everolimus treatment due to oral mucositis | Patients are followed up for 8 weeks after initial enrollment
  Suspension or dose-reduction of everolimus treatment is evaluated by an oncologist
Oral Assessment Guide (Revised) | Patients are followed up for 8 weeks after initial enrollment
  Oral assessment guide is evaluated by a dental/oral surgeon
Health-related quality of life (HRQOL) | Evaluations are executed after the patient enrollment, 4 weeks and the end (8 weeks) of the initiation of the treatment.
  Following QOL questionnaire from (in Japanese) are used for evaluation: FACT-G, GOHAI and SF-36

CONTACTS AND LOCATIONS:
Overall Officials: Akira Yamao, Principal Investigator — Public Health Research Foundation
Locations (1):
- Tokai University, School of Medicine, Isehara, Kanagawa, Japan

REFERENCES:
- [Derived] Nakatsukasa K, Niikura N, Kashiwabara K, Amemiya T, Watanabe KI, Hata H, Kikawa Y, Taniike N, Yamanaka T, Mitsunaga S, Nakagami K, Adachi M, Kondo N, Shibuya Y, Hayashi N, Naito M, Yamashita T, Umeda M, Mukai H, Ota Y. Secondary endpoints analysis in patients with estrogen receptor-positive metastatic breast cancer treated with everolimus and exemestane enrolled in Oral Care-BC. BMC Cancer. 2021 Jan 7;21(1):34. doi: 10.1186/s12885-020-07746-9. PMID 33413212